CLINICAL TRIAL: NCT04429672
Title: Effect of a Socio-educational Intervention on Sexual Health in Young University Students: Randomized Clinical Trial
Brief Title: Effect of a Socio-educational Intervention on Sexual Health in Young University Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Guadalajara (Other)
Collaborators: Universidad de Colima (Other)
Responsible Party: Principal Investigator, Jonathan Josue Vazquez Perez, Principal Investigator, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: VPJJ0001
Record Dates: First submitted 2020-06-07; First posted 2020-06-12 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Sexual Health
MeSH Terms: interventions — Reproductive Physiological Phenomena

STUDY DESIGN:
Intervention Model Description: It is a socio-educational intervention and is composed of five thematic axes; Sexual Rights, Sexuality, Reproductive Health, Sexual Conduct and Life Project divided into ten sessions (two weekly) of 30 minutes each, each session has an established opening, development and closing phase structure
Who Masked: Participant
Masking Description: For the formation of the groups, a restrictive randomization was performed by fixed proportion considering the sample size required for the groups, in which the participant did not identify which group was assigned (simple blind)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (EG) (Experimental): The participants of the Experimental Group receive as treatment the intervention called "The Right to your Sexual Health", which is socio-educational and is composed of five thematic axes; Sexual Rights, Sexuality, Reproductive Health, Sexual Conduct and Life Project divided into ten sessions (two weekly) of 30 minutes each, each session has a structure of the opening, development and closing phase established in a manual for the facilitator, it should be noted that the intervention is applied by a multidisciplinary team in which the areas of medicine, nursing and psychology participate. In addition, Information and Communication Technologies (ICTs) are used through a Moodle platform that has available to participants digital support material as digital presentations on each of the thematic axes, as well as audiovisual material through the Podcast format of conversations concerning each of the axes.
  Interventions: Behavioral: The Right to your Sexual Health
- Control Group (CG) (Active Comparator): The participants of the Control Group receive the usual sexual health intervention applied by Secretary of Health consisting of six sessions (one a week) lasting 50 minutes each using illustrative material through rotating official secretary of health folios on reproductive health, sexually transmitted diseases and sexual violence.
  Interventions: Behavioral: Friendly sexual health services and reproductive for adolescents

INTERVENTIONS:
Behavioral: The Right to your Sexual Health — which is of a socio-educational type and is made up of five thematic axes; Sexual Rights, Sexuality, Reproductive Health, Sexual Behavior and Life Project divided into ten sessions (two weekly) of 30 minutes each, each session has a structure of opening, development and closing phase
  Arms: Experimental Group (EG)
Behavioral: Friendly sexual health services and reproductive for adolescents — consists of six sessions (one a week) lasting 50 minutes each, using illustrative material through official flipcharts of the secretary of health on reproductive health, sexually transmitted diseases and sexual violence
  Arms: Control Group (CG)

SUMMARY:
The sexual health is considered as a state of physical, mental and social well-being in relation to sexuality that requires a positive and respectful approach to sexuality, as well as the possibility of having pleasant and safe sexual experiences, free from all coercion, discrimination and violence. However, lack of family planning, having unprotected sex, unwanted pregnancies, abortions, Sexually Transmitted Infections, lack of acceptance of sexual identity, sexism, having multiple sexual partners and having sex under the influence of alcohol and drugs are some of the main elements that alter the well-being of people's sexual health, especially in the young population. In this sense, different organizations have pointed out the importance of promoting in young people strategies related to providing an adequate level of knowledge in sexual health from a perspective of the exercise of sexual rights to reduce alterations in risky sexual practices and it has been identified that the school environment can be the ideal space for a health services approach to this age group to strengthen their well-being and ensure their development during adulthood. However, the sexual health interventions traditionally implemented by the health services are usually aimed mainly at transmitting knowledge about the benefits of condom use, sexually transmitted diseases and unwanted pregnancies and violence, excluding other elements that make up the sexual health and making use of conventional educational strategies through print media or short educational sessions, which causes little interaction between health personnel and users that consolidates the purpose of the interventions. That said, the implementation of a socio-educational intervention in sexual health that promotes sexual rights, positive attitudes towards sexuality and the prevention of risky sexual behaviors articulated in a model of a life project that motivates them to achieve the ideal stage of life for starting a family in a healthy way through family planning, can promote the strengthening not only of their sexual health but also their well-being for their future development as adults.

ELIGIBILITY:
Inclusion criteria;

* Young college students aged 18 to 24.
* Que reported having an active sex life.
* Who attended the family planning counseling services of the School Clinic.
* Who agreed to participate in the study by signing informed consent.

Exclusion criteria;

* Young people who reported going to private family planning services.
* They were in the gestation stage.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-07-12 (Estimated); Study Completion 2020-12-11 (Estimated)

PRIMARY OUTCOMES:
sexual health | six months
  Changes in the sexual health well-being of young college students. Measuring dimension changes from poor sexual health to good sexual health before and after the intervention, will be measured through proportions and the MacNemar test.

SECONDARY OUTCOMES:
attitudes and opinions towards the sexuality | six months
  Changes in the type of attitudes and opinions towards the sexuality of young university students. Measuring changes in scores obtained from the applicable auto instruments before and after the intervention, is meditated through medians and the Mann-Whitney test.
risky sexual behaviors | six months
  Changes in the type of risky sexual behaviors of young college students. Measuring changes in scores obtained from the applicable auto instruments before and after the intervention, is meditated through medians and the Mann-Whitney test
knowledge and exercise of the sexual rights | six months
  Changes in the knowledge and exercise of the sexual rights of young university students. Measuring changes in scores obtained from the applicable auto instruments before and after the intervention, it is meditated through medians and the Mann-Whitney test.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan J Vazquez Perez, Msc, Principal Investigator — University of Guadalajara; Benjamin Trujillo Hernández, Dsc, Study Director — Universidad de Colima; José C Vásquez Jiménez, Dsc, Study Director — Universidad de Colima
Locations (1):
- Southern University Center, Zapotlán el Grande, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Villalobos A, Castro F, Rojas R, Allen B. [Contraception in Mexican adolescents in upper secondary schools: use and unmet needs]. Salud Publica Mex. 2017 Sep-Oct;59(5):566-576. doi: 10.21149/8481. Spanish. PMID 29267654